CLINICAL TRIAL: NCT01137292
Title: Voriconazole In High-Risk Patients With Invasive Fungal Infections In Slovakia. An Open, Prospective, Non-Comparative Study
Brief Title: Open, Non Comparative Study Of Voriconazole In Slovak Patients With Very High Risk Of Developing An Invasive Fungal Infection
Acronym: Ve-RIFI
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501082
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Invasive Fungal Infections
Keywords: observational study; voriconazole; high-risk patients
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Active Treatment: Patients who are eligible for voriconazole treatment according to their physician decision.
  Interventions: Drug: voriconazole (VFEND®)

INTERVENTIONS:
Drug: voriconazole (VFEND®) — The use and dosage recommendations for voriconazole (VFEND®) will take place on the basis of the Summary of Product Characteristics (SmPC) and will be adjusted solely according to medical and therapeutic necessity. The formulation and dose will be managed by the treating physician according to the SmPC, disease and clinical situation. According to the SmPC, in the adults the treatment should be started with the loading dose of 6 mg/kg of voriconazole iv. every 12 hours (during the first 24 hrs) followed by the maintenance dose of 4 mg/kg BID. For peroral formulations, the initial dose should be depending on the weight of the patient 400 mg or 200 mg BID during the first 24 hrs, followed by the maintenance dose of 200 mg or 100 mg of voriconazole BID respectively For paediatric population (<12 years of age), there is no initial dose necessary. Depending on the formulation, the daily dosage should be in children 7 mg/kg iv. BID or 200 mg of voriconazole orally BID.

SUMMARY:
Assessment of safety and efficacy of voriconazole in real-life setting in the treatment of high risk patients with invasive fungal infections. The study is conducted in Slovakia only.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of age 2 years or older.
* High-risk patients with proven, probable or possible invasive fungal infection (IFI) according to the EORTC/MSG criteria.
* Patients indicated for secondary prophylaxis of invasive aspergillosis.

Exclusion Criteria:

* Patients with known hypersensitivity to voriconazole or to any of the excipients.
* Patients with contraindicated concomitant medications according to the SmPC.
* Children less than 2 years of age.
* Pregnancy and lactation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients older than 2 years with invasive fungal infections.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501082&StudyName=Open%2C%20Non%20Comparative%20Study%20Of%20Voriconazole%20In%20Slovak%20Patients%20With%20Very%20High%20Risk%20Of%20Developing%20An%20Invasive%20Fungal%20Infection

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole: In adults, treatment was started with the loading dose of 6 mg/kg of voriconazole intravenously every 12 hours (during the first 24 hrs) followed by the maintenance dose of 4 mg/kg twice a day (BID). Adults with a weight of >40 kg receiving the oral formulation received a loading dose of 400 mg BID during the first 24 hours, followed by a maintenance dose of 200 mg BID for the duration of the study.
  Adults with a weight of <40 kg receiving the oral formulation received a loading dose of 200 mg BID during the first 24 hours, followed by a maintenance dose of 100 mg BID for the duration of the study. Pediatric participants under 12 years of age received 7 mg/kg IV BID or 200 mg orally BID for the duration of the study. A loading dose was not required in participants under 12 years of age.
Period: Overall Study
Arm/Group | Voriconazole
Started | 177
Completed | 123
Not Completed | 54
Not completed — Death | 30
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 13
Not completed — Lost to Follow-up | 1
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole
Number analyzed (Participants) | 177
Age, Customized [Number; unit: participants]
  < 2 years | 3
  2 to 18 years | 16
  19 to 44 years | 52
  45 to 64 years | 80
  > = 65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 104
Number of Participants Having Certain Methods of Diagnosis of Invasive Aspergillosis [Number; unit: participants]
  Hi-Resolution Computed Tomography | 91
  Galactomannan | 55
  Polymerase Chain Reaction (PCR) | 5
  Blood Culture | 8
  Bronchoalveolar Lavage (BAL) | 23
  Biopsy | 2
Number of Participants with Risk Factors of Invasive Fungal Infections [Number; unit: participants]
  Radiotherapy | 8
  Neuropenia | 104
  Autologic Bone Marrow Transplant | 11
  Polytrauma | 13
  Antibiotic Prophylaxis | 81
  Immunosuppressive Treatment | 42
  Graft-Versus-Host Disease | 7
  Malignant Tumour | 110
  Chemotherapy | 122
  Undergone Surgery | 23
  Central Venous Catether | 110
  Ventilation (Intubation) | 32
  Hemodialysis | 5
  Antifungal Prophylaxis | 114
  Primary/Secondary Immunodeficiency | 101
  Total Parental Nutrition | 35
  Cytomegalovirus Infection | 13
  Allogenic Bone Marrow Transplant | 13
  Diabetes Mellitus | 10
  Organ Transplant | 3
  Previous Antibiotic Treatment | 120
  Steroid Treatment | 74
  Mucositisis | 38
  Other Invasive Mycosis | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical and/or Mycological Efficacy by Response at the End of Treatment (EOT) Visit
Description: Clinical, mycological responses: clinical cure, clinical improvement, no clinical cure, mycological cure, no mycological cure, and no mycological culture performed. Participants could have had more than one response. Responses were based on the investigator's judgement according to the Infectious Disease Society of America, European Conference on Infections in Leukemia, and European Committee on Antimicrobial Susceptibility Testing guidelines.
Time Frame: up to 2 weeks (EOT visit)
Population: Full Analysis Set (FAS) = all enrolled participants who were administered the study medication and had post baseline documentation of efficacy available.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 177
participants
  Clinical Cure | 64
  Clinical Improvement | 64
  No Clinical Cure | 36
  Mycological Cure | 34
  No Mycological Cure | 10
  No Mycological Culture Performed | 40

2. Primary Outcome: Number of Participants With Clinical and/or Mycological Efficacy by Response at the Test-of-Cure Visit
Description: Clinical, mycological responses: clinical cure, clinical improvement, no clinical cure, mycological cure, no mycological cure, no mycological culture performed, death, and lost from follow-up. Participants could have had more than one response. Responses were based on the investigator's judgement according to the Infectious Disease Society of America, European Conference on Infections in Leukemia, and European Committee on Antimicrobial Susceptibility Testing guidelines.
Time Frame: more than 2 weeks (Test-of-Cure visit)
Population: FAS.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 177
participants
  Clinical Cure | 54
  Clinical Improvement | 46
  No Clinical Cure | 7
  Mycological Cure | 31
  No Mycological Cure | 1
  No Mycological Culture Performed | 19
  Death | 41
  Lost From Follow-Up | 11

3. Primary Outcome: Number of Participants With Investigator's Satisfaction With the Efficacy of Voriconazole Assessment at the EOT Visit
Description: Investigator's Satisfaction Responses: very good, good, moderate, poor. Responses were based on the investigator's judgement.
Time Frame: up to 2 weeks (EOT visit)
Population: FAS. Number or participants analyzed = Number of participants with Investigator's satisfaction response for the efficacy of voriconazole at the EOT Visit.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 172
participants
  Very Good | 85
  Good | 49
  Moderate | 33
  Poor | 5

4. Primary Outcome: Number of Participants With Investigator's Satisfaction With the Tolerability of Voriconazole Assessment at the EOT Visit
Description: as for outcome 3
Time Frame: up to 2 weeks (EOT visit)
Population: FAS. Number or participants analyzed = Number of participants with Investigator's satisfaction response for the tolerability of voriconazole at the EOT Visit.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 174
participants
  Very Good | 105
  Good | 61
  Moderate | 8
  Poor | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Voriconazole
Serious Adverse Events (participants affected / at risk) | 34/177
Other Adverse Events (participants affected / at risk) | 6/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=177)
Bone marrow disorder (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 5
Cardiopulmonary failure (Cardiac disorders) | 4
Disease progression (General disorders) | 1
Multi-organ failure (General disorders) | 8
Sudden death (General disorders) | 1
Aspergillosis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 2
Multiple injuries (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage intracranial (Nervous system disorders) | 3
Haemorrhagic stroke (Nervous system disorders) | 1
Locked-in syndrome (Nervous system disorders) | 1
Crush syndrome (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=177)
Liver disorder (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acrodermatitis (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Hypertensive crisis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.